CLINICAL TRIAL: NCT02977494
Title: Daratumumab in Combination With Bortezomib and Dexamethasone in Subjects With Relapsed or Relapsed and Refractory Multiple Myeloma and Severe Renal Impairment Including Subjects Undergoing Hemodialysis: A Phase 2, Open-label, Multicenter Trial
Brief Title: Daratumumab in Combination With Bortezomib and Dexamethasone in Subjects With Relapsed or Relapsed and Refractory Multiple Myeloma and Severe Renal Impairment
Acronym: GMMG-DANTE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-000433-51
Record Dates: First submitted 2016-11-17; First posted 2016-11-30 (Estimated); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab; Bortezomib; Dexamethasone; dexamethasone acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Daratumumab Bortezomib (Experimental)
  Interventions: Drug: Daratumumab; Drug: Bortezomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Daratumumab — Daratumumab (JNJ-54767414) is a novel human IgG1monoclonal Antibody (mAb) that binds with high affinity to a unique epitope on CD38
  Other Names: Darzalex
Drug: Bortezomib
  Other Names: Velcade
Drug: Dexamethasone
  Other Names: Fortecortin

SUMMARY:
Myeloma patients with renal impairment need a rapid and effective reduction of tumor burden to enable renal recovery, which is correlated with prognosis of the patients. However, effective combination regimens are often hampered by necessary dose reductions or increased toxicity in renally impaired patients. The well known positive effects on renal impairment by Bortezomib combined with Daratumumab, which, as all monoclonal Antibody, is not renally excreted or metabolized and as so far known should not add significant toxicity but efficacy, makes the proposed combination of Daratumumab, Bortezomib and Dexamethasone highly attractive for renally impaired MM patients.

In the current clinical trials with Daratumumab patients with renal function impairment (GFR ≤ 20 ml/min) were so far excluded. Consequently questions about efficacy, safety and pharmacokinetics of Daratumumab in combination with Bortezomib and Dexamethasone in patients with relapsed and refractory MM and severe renal impairment are still unanswered. This trial will answer these questions for a patient group, who has still an unmet need for novel and effective treatment options

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be at least 18 years of age
2. Written informed consent
3. Subjects must have had documented multiple myeloma requiring treatment as defined by the criteria below:

   Monoclonal plasma cells in the bone marrow > 10% and/or presence of a biopsy-proven plasmacytoma at some point in their disease history requiring treatment according diagnostic criteria (IMWG updated criteria 2014, Rajkumar et al. 2014) see appendix I With measurable disease at screening (serum M-protein > 500 mg/dl or urine M-protein > 200 mg/24h, in case of oligosecretory MM serum free light chain > 10 mg/dl and abnormal kappa/lambda free light chain ratio)
4. GFR < 30 ml/min and /or subjects undergoing hemodialysis
5. Subject must have received at least 1 prior treatment line
6. Subjects must have documented evidence of progressive disease after the last treatment line
7. ECOG performance status 0-3 (ECOG 3 is only allowed if due to myeloma disease)
8. Subjects must have certain pretreatment laboratory values meeting the following criteria during the Screening Phase:

   1. Hemoglobin ≥7.5 g/dl (4,66 mmol/L; prior red blood cells (RBC) transfusion or recombinant human erythropoietin use is permitted).
   2. Absolute neutrophil count ≥ 1.0 x109/L (granulocyte colony stimulating factor (GCSF) use is permitted);
   3. Platelet count more or equal 70 x109/L for subjects in whom ˂ 50% of bone marrow nucleated cells are plasma cells; otherwise platelet count ˃ 50 x 109/L (transfusions are not permitted to achieve this minimum platelet count ),
   4. Aspartate aminotransferase (AST) ≤ 2,5 x upper limit of normal (ULN);
   5. Alanine aminotransferase (ALT) ≤ 2,5 x ULN
   6. Total bilirubin ≤ 2.0 x ULN ,except in subjects with congenital bilirubinemia, such as Gilbert syndrome (direct bilirubin ≤ 2.0 x ULN
   7. Corrected serum calcium ≤ 14 mg/dl (≤3,5mmol/L); or free ionized calcium ˂ 6,5 mg/dL(˂1,6 mmol/L)
9. Women of childbearing potential must commit to either abstain continuously from heterosexual sexual intercourse or to use 2 methods of reliable birth control simultaneously. This includes one highly effective form of contraception (tubal ligation, intrauterine device [IUD], hormonal [birth control pills, injections, hormonal patches, vaginal rings or implants] or partner's vasectomy) and one additional effective contraceptive method (male latex or synthetic condom, diaphragm, or cervical cap). Contraception must begin 4 weeks prior to dosing. Reliable contraception is indicated even where there has been a history of infertility, unless due to hysterectomy.
10. A woman of childbearing potential must have a negative urine or serum pregnancy test at screening within 14 days prior to treatment start.

Exclusion Criteria:

1. Subject has received prior Daratumumab or other Anti-CD38 antibodies (previous treatment with Elotuzumab is allowed)
2. Evidence of intolerance to bortezomib or known allergies, hypersensitivity or intolerance to monoclonal antibodies
3. Subject has received anti-myeloma treatment within 2 weeks of Cycle 1, day 1. The only exception is emergency use of a short course of corticosteroids (equivalent of Dexamethasone 40 mg/day for a maximum of 4 days) before treatment.
4. Active graft-versus host disease under immunosuppressive treatment
5. Subject is a woman who is pregnant or breastfeeding
6. Prior invasive malignancy within 5 years before trial inclusion
7. Active, uncontrolled infection.
8. Subject has peripheral neuropathy ≥ 3 or neuropathic pain Grade 2 or higher
9. Subject has either of the following:

   1. Known chronic obstructive pulmonary disease (COPD) with a forced expiratory volume in 1 second (FEV1) <50% of predicted normal. Note that FEV1 testing is only required for subjects suspected of having COPD
   2. Known moderate or severe persistent asthma, or currently has uncontrolled asthma of any classification. (Note that subjects who currently have controlled intermittent asthma or controlled mild persistent asthma are allowed to participate in the study).
10. Subject has clinically significant cardiac disease, including myocardial infarction within 6 months before date of study entry, unstable angina, cardiac insufficiency New York Heart Association (NYHA) Class III-IV or uncontrolled arrhythmia
11. Subject has a diagnosis of primary amyloidosis, monoclonal gammopathy of undetermined significance, or smoldering multiple myeloma. Monoclonal gammopathy of undetermined significant is defined by presence of serum M-protein ˂ 3 g/dL; absence of lytic bone lesions, anemia, hypercalcemia and renal insufficiency related to M-protein; and (if determined) proportion of plasma cells in the bone marrow of 10% or less (Kyle et al. 2003). Smoldering multiple myeloma is defined as asymptomatic multiple myeloma with absence of related organ or tissue impairment and organ damage (Kyle et al., 2003, 2007).
12. Subject has a diagnosis of Waldenström's disease, or other conditions in which IgM M-protein is present in the absence of a clonal plasma cell infiltration with lytic bone lesions.
13. Subject has had radiation therapy within 14 days of treatment
14. Subject has had plasmapheresis within 14 days of treatment. Screening laboratory values have to be performed after end of plasmapheresis.
15. Subject is known to be seropositive for human immunodeficiency virus (HIV) or hepatitis B (defined by a positive test for hepatitis B surface antigen (HBsAg) or antibodies to hepatitis B surface and core antigen (anti HBs and anti HBc respectively), or hepatitis C (anti-HCV antibody positive or HCV RNA quantitation positive).
16. Subject has had major surgery within 2 weeks before treatment und has not fully recovered from surgery, or has surgery panned during the time the subject is expected to participate in the study.
17. Incidence of gastrointestinal disease that may significantly alter the absorption of oral drugs
18. Subject has any concurrent medical or psychiatric condition or disease (eg. active systemic infection, uncontrolled diabetes, acute diffuse infiltrative pulmonary disease) that is likely to interfere with the study procedures or results, or that in the opinion of the investigator, would constitute a hazard for the participating in this study.
19. Subject has known allergies, hypersensitivity, or intolerance to corticosteroids, monoclonal antibodies or human proteins, or their excipients (refer to respective package inserts or Investigator's Brochure), or known sensitivity to mammalian-derived products.
20. Subject is known or suspected of not being able to comply with the study protocol (eg. because of alcoholism, drug dependency, or psychological disorder). Subject has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the subject (eg, compromise the well-being) or that could prevent, limit or confound the protocol-specified assessments. Subject is taking any prohibited medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2021-06 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficacy (overall response rate, ORR according to IMWG recommendations) of the combination of daratumumab, bortezomib and dexamethasone in subjects with relapsed and refractory MM and impaired renal function | two years

CONTACTS AND LOCATIONS:
Locations (10):
- Germany (9):
  - Charité Universitätsmedizin BerlinCampus Benjamin Franklin, Berlin
  - Vivantes Klinikum Neukölln, Berlin
  - Klinikum Chemnitz GmbH, Chemnitz
  - Katholische Karl-Leisner Klinikum Goch, Goch
  - Asklepios Klinik Altona, Hamburg
  - University Hospital Hamburg Eppendorf, Hamburg
  - Universitätsklinikum Heidelberg, Heidelberg
  - Univerisity Hospital Muenster, Münster
  - University Hospital, Tübingen
- Alexandra Hopsital, Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided